CLINICAL TRIAL: NCT04371055
Title: Intensive Heart Rhythm Monitoring to Decrease Ischemic Stroke and Systemic Embolism - the Find-AF 2 Study
Brief Title: Intensive Rhythm Monitoring to Decrease Ischemic Stroke and Systemic Embolism - the Find-AF 2 Study
Acronym: Find-AF2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Rolf Wachter, Professor for Clinical and Interventional Cardiology, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Find-AF 2
Record Dates: First submitted 2020-04-24; First posted 2020-05-01 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Stroke; Atrial Fibrillation
Keywords: Atrial Fibrillation; Ischemic Stroke; ECG Monitoring; Secondary Prevention
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomised, parallel, multicenter interventional trial with blinded assessment of the primary endpoint
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risk-adapted ECG monitoring for atrial fibrillation (Experimental): Intervention Group with high Risk for AF:
  Continuous Rhythm Monitoring using an implantable cardiac Monitor
  Intervention group with low risk for AF:
  7-day Holter ECG at baseline, after 3 and 12 months and then annually until the end of the study or the first occurrence of atrial Fibrillation
  Interventions: Other: 7-day Holter ECG; Other: Implantable cardiac monitor
- Standard of Care (Other): Standard of care rhythm monitoring
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: 7-day Holter ECG — 7-day Holter ECG at baseline and after 3 and 12 months and then annually until the end of the study or the first (in patients with low risk of atrial fibrillation)
  Arms: Risk-adapted ECG monitoring for atrial fibrillation
Other: Implantable cardiac monitor — Continuous rhythm monitoring using an implantable cardiac monitor
  Arms: Risk-adapted ECG monitoring for atrial fibrillation
Other: Standard of care — Usual care according to current guidelines (in patients with low and high risk of atrial fibrillation)
  Arms: Standard of Care

SUMMARY:
Patients who have suffered a stroke are having an increased risk of having recurrent stroke in the future. This risk of stroke is increased by atrial fibrillation, which often "comes and goes" (called paroxysmal) and hence escapes routine diagnostics. The hypothesis of Find-AF 2 is that enhanced (evaluation in a ECG core lab), prolonged (at least 7 days of rhythm monitoring annually) and intensified (continuous rhythm monitoring in high risk patients) not only finds atrial fibrillation more often, but that changes in therapeutic management (e. g. start of anticoagulation after detection of atrial fibrillation) results in a decrease of cardioembolism (which can be either recurrent stroke or systemic embolism).

To prove this hypothesis, patients will be randomised into two groups: the first group will receive the currently available standard care for patients with stroke. In the second group, cardiac rhythm monitoring adapted to the risk of the occurrence of atrial fibrillation is performed - either with a 7-day long-term ECG (at baseline, after 3 and 12 months and every 12 months thereafter) or with continuous monitoring using an implantable cardiac monitor. If atrial fibrillation is detected, this information will be given to the treating study physician. Any therapeutic decision is at the discretion of the treating physician, but should follow current guidelines.

DETAILED DESCRIPTION:
The Find AF 2 study will investigate whether intensified rhythm monitoring in patients with recent ischemic stroke leads to a decrease in recurrent thromboembolism (defined as recurrent ischemic stroke or systemic embolism). This will be achieved by identifying patients with paroxysmal atrial fibrillation and subsequently switching secondary prevention therapy from antiplatelet therapy to oral anticoagulation. The intensity of heart rhythm monitoring will be risk-adjusted: Patients with an estimated low risk of atrial fibrillation receive a 7-day Holter ECG, which is repeated after 3 and 12 months and annually thereafter. Patients with a high risk of atrial fibrillation (defined by increased supraventricular ectopic activity) receive continuous ECG monitoring using an implanted loop recorder. The control arm is treated according to local standards, which includes cardiac rhythm monitoring for at least 24 hours according to current guidelines. Prior to randomization, a 24-hour Holter ECG is performed in both study arms, ensuring minimal ECG monitoring for patients in the control arm and allowing risk stratification in the intervention arm. Additional ECG monitoring using stroke telemetry and/or additional Holter ECGs is possible according to local standards, provided it does not exceed 7 days. Patients in both study arms will be followed up for at least 24 months.

It should be noted that this study only provides diagnostic information, the therapeutic decision is left to the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Recent ischemic stroke (sudden focal neurologic deficit lasting > 24h consistent with the territory of a major cerebral artery) and/or a corresponding lesion on brain imaging within the last 30 days
2. Age ≥ 60 years
3. Patient without or with only slight disability (modified Rankin Scale score ≤ 2) before onset of stroke-related symptoms.
4. Written informed consent

Exclusion Criteria:

1. Known history of atrial fibrillation/flutter or atrial fibrillation/flutter on admission ECG
2. Current indication or contraindication for oral anticoagulation at randomisation
3. Intracerebral bleeding in medical history
4. Patient scheduled for ECG-monitoring lasting > 7 days (Holter-ECG, implanted loop recorder, etc.)
5. Implanted pacemaker device or cardioverter/ defibrillator
6. Patient not willing to be treated with oral anticoagulants
7. Carotid artery stenosis ipsilateral to the current ischemic stroke needing operation or intervention.
8. History of carotid endarterectomy or percutaneous intervention of cerebral artery within the last 30 days.
9. Life expectancy <1 year for reasons other than stroke (e.g. metastatic cancer)
10. patients under legal supervision or guardianship
11. psychological/mental or other inabilities to supply required information (e.g. fill out the questionnaire due to dementia, language difficulties,...) or participate in the required tests
12. participation in other randomised interventional trials
13. suspected lack of compliance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5227 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Time until recurrent ischemic stroke or systemic embolism | from the date of randomization until the date of first documented ischemic stroke or date of first systemic embolism, whichever comes first, assessed up to 60 months
  The trial will be event driven. The minimum follow-up in each patient is 24 months, but may be followed for up to 60 months.
Primary safety endpoint: Time until the first haemorrhagic stroke | from the date of randomization until the date of first documented haemorrhagic stroke, assessed up to 60 months
  Time until the first haemorrhagic stroke

SECONDARY OUTCOMES:
Time until the combination of stroke, myocardial infarction and cardiovascular death | from the date of randomization until the date of first documented stroke, the date of myocardial infarction and the date of cardiovascular death, whichever comes first, assessed up to 60 months
  Time until the combination of stroke, myocardial infarction and cardiovascular death
Time until any stroke | from the date of randomization until the date of first documented any stroke, assessed up to 60 months
  Time until any stroke
Time until new onset of AF | from the date of randomization until the date of first documented AF, assessed up to 60 months
  Time until new onset of Atrial Fibrillation
Time until all cause mortality | from the date of randomization until the date of all cause mortality assessed up to 60 months
  Time until all cause mortality
Time until myocardial infarction | from the date of randomization until the date of all myocardial infarction, assessed up to 60 months
  Time until myocardial infarction
Changes in quality of life (QoL), measured by the stroke impact scale (SIS-16) | Mean change from baseline until study end assessed up to 60 months in both study arms
  Changes in quality of life (QoL), measured by the stroke impact scale (SIS-16). The SIS-16 ranges from 16 to 80, with higher scores showing better Quality of life.
Changes in the EQ-5D five dimensional Quality of Life (QoL) | Mean change from baseline until study end assessed up to 60 months in both study arms
  Changes in the EQ-5D five dimensional Quality of Life (QoL)
Changes in the overall QoL visual analog scale | Mean change from baseline until study end assessed up to 60 months in both study arms, ranging from 0 to 100, with higher values indicating better quality of life
  Changes in the overall QoL visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Wachter, Prof. Dr., Study Chair — University of Leipzig, Clinic and Policlinis for Cardiology; Klaus Gröschel, Prof. Dr., Principal Investigator — University of Mainz, Clinic and Policlinis for Neurology
Locations (52):
- Germany (52):
  - ISD München, München, Bavaria
  - Klinikum Nürnberg, Nuremberg, Bavaria
  - Klinikum Bremen Mitte, Bremen, City state Bremen
  - University of Leipzig, Clinic for Neurology, Leipzig, Saxony
  - Vivantes Klinikum Neukölln Berlin, Berlin, State of Berlin
  - Klinikum Altenburger Land, Altenburg
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg
  - Universitätsklinikum Augsburg, Augsburg
  - Rhön Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale
  - Sozialstiftung Bamberg; Klinikum am Bruderwald, Bamberg
  - BG Klinikum, Unfall-KH Berlin gGmbH, Berlin
  - Vivantes, Humboldt-Klinikum Berlin, Berlin
  - Vivantes Klinikum Spandau, Berlin-Spandau
  - Evangelisches Klinikum Bethel, Klinik für Neurologie, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Coburg, Medizinische Klinik für Innere Medizin und Kardiologie, Coburg
  - Klinikum Darmstadt, Darmstadt
  - Städtisches Klinikum Dresden, Standort Friedrichstadt, Dresden
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - University of Essen, Clinic for Neurology, Essen
  - Klinikum Frankfurt Höchst, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Klinikum Fulda, Fulda
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - University of Göttingen, Clinic for Neurology, Göttingen
  - Bezirkskrankenhaus Günzburg, Günzburg
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Albertinenkrankenhaus Hamburg, Hamburg
  - Asklepios Klinik Altona Hamburg, Hamburg
  - Asklepios Klinik Wandsbek, Hamburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Höxter, Höxter
  - Klinikum Ibbenbüren, Ibbenbueren
  - Klinikum St. Georg Leipzig, Leipzig
  - Städtisches Klinikum Lüneburg gemeinnützige GmbH, Lüneburg
  - University of Mainz, Clinic for Neurology, Mainz
  - Carl-von-Basedow Klinikum Merseburg, Merseburg
  - Klinikum Minden, Minden
  - Ökumenisches Hainich Klinikum Mühlhausen, Mühlhausen
  - Universitätsklinikum Münster, Münster
  - Klinikum Osnabrück GmbH, Osnabrück
  - Klinikum Passau, Passau
  - Nordwest-Krankenhaus Sanderbusch, Klinik für Neurologie, Sande
  - Kreisklinikum Siegen, Siegen
  - Kliniken Südostbayern AG, Klinikum Traunstein, Traunstein
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Helios Dr. Horst Schmidt-Kliniken Wiesbaden, Wiesbaden
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after publication of the major results

REFERENCES:
- [Background] Uhe T, Wasser K, Weber-Kruger M, Schabitz WR, Kohrmann M, Brachmann J, Laufs U, Dichgans M, Gelbrich G, Petroff D, Prettin C, Michalski D, Kraft A, Etgen T, Schellinger PD, Soda H, Bethke F, Ertl M, Kallmunzer B, Grond M, Althaus K, Hamann GF, Mende M, Wagner M, Groschel S, Uphaus T, Groschel K, Wachter R; Find-AF 2 study group. Intensive heart rhythm monitoring to decrease ischemic stroke and systemic embolism-the Find-AF 2 study-rationale and design. Am Heart J. 2023 Nov;265:66-76. doi: 10.1016/j.ahj.2023.06.016. Epub 2023 Jul 7. PMID 37422010
- [Derived] Wasser K, Uhe T, Schabitz WR, Kohrmann M, Dichgans M, Brachmann J, Laufs U, Gelbrich G, Petroff D, Prettin C, Michalski D, Pelz J, Kraft A, Etgen T, Soda H, Bethke F, Schellinger PD, Althaus K, Hamann GF, Grond M, Kallmunzer B, Petersen M, Pallesen LP, Ertl M, Zickler P, Poli S, Haeusler KG, Steiner T, Sparenberg P, Kermer P, Kopczak A, Kellert L, Nuckel M, Liman J, Ringleb PA, Mende M, Wagner M, Bochert D, Schnieder M, Amanzada I, Groschel S, Hahn M, Uphaus T, Groschel K, Wachter R; Find-AF 2 study group. Baseline characteristics of patients with acute ischaemic stroke included in the randomised controlled Find-AF 2 trial. Neurol Res Pract. 2025 Jun 26;7(1):45. doi: 10.1186/s42466-025-00399-8. PMID 40571918
- See also: Study homepage with information for medical experts and the general public — http://www.find-af2.com